CLINICAL TRIAL: NCT02689427
Title: A Phase IIB Study of Neoadjuvant ZT Regimen (Enzalutamide Therapy in Combination With Weekly Paclitaxel) for Androgen Receptor (AR)-Positive Triple-Negative Breast Cancer
Brief Title: Enzalutamide and Paclitaxel Before Surgery in Treating Patients With Stage I-III Androgen Receptor-Positive Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0488; NCI-2016-00367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0488 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Invasive Breast Carcinoma; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
Keywords: Androgen Receptor positive TNBC
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — enzalutamide; Sentinel Lymph Node Biopsy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzalutamide, paclitaxel) (Experimental): Patients receive enzalutamide PO daily on days 1-7 and paclitaxel IV over 2 hours on day 1. Treatments repeat every 7 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  SURGERY: After 12 cycles of therapy, patients undergo surgical resection of primary tumor with or without lymph node biopsy or complete axillary dissection.
  Interventions: Procedure: Axillary Lymph Node Dissection; Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Procedure: Lymph Node Biopsy; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Axillary Lymph Node Dissection — Undergo axillary lymph node dissection
  Other Names: ALND; Axillary Dissection; Axillary Lymphadenectomy; Axillary Node Dissection; Excision Axillary Lymph Nodes
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Lymph Node Biopsy — Undergo lymph node biopsy
  Other Names: Biopsy of Lymph Node
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection of primary tumor

SUMMARY:
This phase IIB trial studies how well enzalutamide and paclitaxel before surgery works in treating patients with stage I-III androgen receptor-positive triple-negative breast cancer. Androgens can cause the growth of triple-negative breast cancer. Anti-hormone therapy, such as enzalutamide, prevent androgen from binding to the androgen receptor, thereby decreasing cell growth and causing tumor cell death. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving enzalutamide and paclitaxel before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. This treatment study is part of the MD Anderson Moonshot initiative.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the pathologic complete response (pCR) and residual cancer burden-index (RCB-I) rates of patients with triple-negative breast cancer (TNBC) who were non-responders to initial anthracycline and cyclophosphamide chemotherapy and who were treated with enzalutamide in combination with weekly paclitaxel in the neoadjuvant setting.

SECONDARY OBJECTIVES:

I. To estimate progression free survival (PFS) distribution of androgen receptor (AR)-positive TNBC patients who were nonresponders to initial anthracycline and cyclophosphamide chemotherapy, treated with enzalutamide in combination with weekly paclitaxel in the neoadjuvant setting.

II. To determine the safety of administering enzalutamide in combination with weekly paclitaxel in the neoadjuvant setting.

EXPLORATORY OBJECTIVES:

I. To investigate the association between biomarkers in the peripheral blood and tumor tissue with safety and efficacy for TNBC patients who were treated with enzalutamide and treatment in combination with weekly paclitaxel in the neoadjuvant setting.

II. To investigate the correlation between circulating tumor cells (CTC) characteristics and/or gene profiles and treatment response of enzalutamide and taxane.

OUTLINE:

Patients receive enzalutamide orally (PO) daily on days 1-7 and paclitaxel intravenously (IV) over 2 hours on day 1. Treatments repeat every 7 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

SURGERY: After 12 cycles of therapy, patients undergo surgical resection of primary tumor with or without lymph node biopsy or complete axillary dissection.

After completion of study treatment, patients are followed up within 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Patients with histologically confirmed intact primary cancer that is confirmed invasive carcinoma of the breast, with at least 1.0 cm residual disease as measured by mammography, ultrasound, or breast MRI after neoadjuvant anthracycline based chemotherapy.
3. Triple-negative breast cancer defined as ER<10%; PR<10% by immunohistochemistry (IHC) and HER2 0-1+ by IHC, or 2+ FISH non-amplified.
4. Androgen Receptor will be quantified using CLIA-compliant assays for AR on a biopsy specimen obtained prior to initiation of treatment.. AR-positivity is defined as > 10% of nuclear staining.
5. AJCC 7th edition stage I-III Breast Cancer
6. Men or women 18 years of age or older.
7. Patients must have a performance status of (0-1) on the ECOG performance scale
8. Negative serum or urine pregnancy test must be done within 72 hours before the first dose of the study medication for women of childbearing potential as per institutional guidelines. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo pregnancy test.
9. Men on study must use a condom if having sex with a pregnant woman.
10. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration
11. Patient must have adequate organ function as determined by the following laboratory values:

    * Absolute neutrophil count ≥ 1,500 /μL
    * Platelets ≥ 100,000 / μL
    * Hemoglobin ≥ 9 g/dL
    * Creatinine Clearance > 50 ml/min
    * Total Bilirubin < 1.5 x ULN
    * ALT/AST < 2.5 x ULN

Exclusion Criteria:

1. Patients who have received any previous antitumor therapies (other than anthracyclinebased neoadjuvant chemotherapy for the current cancer event).
2. Female patients must not be breast-feeding at screening or planning to become pregnant during the course of therapy.
3. Patients having major surgery within 21 days before Cycle 1, Day 1.
4. Patients with known history of hypersensitivity to paclitaxel that did not resolve with pre- medication.
5. Patients with left ventricular ejection fraction <50% or 10% decrease from baseline on echocardiogram after anthracycline based chemotherapy.
6. Patients with gastrointestinal impairment that would affect the absorption of Enzalutamide; or previous history of colitis.
7. Subjects requiring daily corticosteroids, other than those given as premedication for the anthracycline-based chemotherapy.
8. Patients with known or suspected brain metastasis or active leptomeningeal disease.
9. History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma) at any time in the past. Also, history of loss of consciousness or transient ischemic attack within 12 months of Day 1 visit.
10. Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide + Paclitaxel: Patients receive 120mg enzalutamide PO daily on days 1-7 and paclitaxel IV over 2 hours on day 1. Treatments repeat every 7 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Enzalutamide + Paclitaxel
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide + Paclitaxel
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: Years] | 57.5 [39 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: RCB Status
Description: The RCB (Residual Cancer Burden) is a continuous variable derived from the primary tumor dimensions, cellularity of the tumor bed, and axillary nodal burden. RCB can be divided into four classes (RCB-0 to RCB-III) and will be collected as part of the study. RCB-0 (pCR), Minimal RCB (RCB-I), Moderate RCB (RCB-II), and Extensive RCB (RCB-III)
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide + Paclitaxel
Number analyzed (Participants) | 24
Participants
  pcR | 4
  RCB-I | 6
  RCB-II | 8
  RCB-III | 6

2. Primary Outcome: Incidence of Residual Cancer Burden-index
Description: Using a Simon optimal two-stage design with alpha = beta = 10%, and then setting the threshold for an acceptable pathologic complete response or residual cancer burden-index rate at 20%. Will be estimated by the proportion of patients with pathologic complete response (residual cancer burden-zero) or residual cancer burden-index as the response rate along with an appropriate 95% confidence interval.
Time Frame: Up to 30 days after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival Distribution
Description: Estimated using Kaplan-Meier method. Progression of disease defined as > 20% increase in tumor.
Time Frame: From enrollment to progression of disease or death whichever comes first, up to 30 days after surgery
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Levels of Biomarkers of Response
Description: Correlated with pathologic response to treatment using appropriate statistical analyses for the biomarker of interest.
Time Frame: Up to 30 days after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Enzalutamide + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Paclitaxel (N=24)
Cholecystitis (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Paclitaxel (N=24)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Neutrophil Count decreased (Investigations) | 9 (12)
Anemia (Blood and lymphatic system disorders) | 8 (15)
Peripheral Sensory Neuropathy (Nervous system disorders) | 8 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Fatigue (General disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02689427/Prot_SAP_000.pdf